CLINICAL TRIAL: NCT00010153
Title: A Double-Blind Phase III Clinical Trial to Compare the Effects of a Pre-Operatively Administered Single Dose of "Faslodex" (Long-Acting ICI 182.780) With Placebo on Tumor Recurrence in Pre- and Postmenopausal Women Treated for Operable First Primary Breast Cancer
Brief Title: ICI 182780 in Treating Women With Stage I or Stage II Primary Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Breast International Group (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-10963; EORTC-10963; BIG-EORTC-10963
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

INTERVENTIONS:
Drug: fulvestrant
Procedure: conventional surgery

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using ICI 182780 before surgery may block the uptake of estrogen by the tumor cells and prevent metastases. It is not yet known if ICI 182780 is effective in preventing breast cancer metastases.

PURPOSE: Randomized phase III trial to study the effectiveness of ICI 182780 given before surgery in treating women who have stage I or stage II primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the inhibitory effect of ICI 182780 on the development of metastasis, as measured by disease-free survival and overall survival, in women with operable stage I or II primary breast cancer.
* Determine toxicity of this regimen in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center and menopausal status (premenopausal vs postmenopausal).

Patients are randomized to receive either ICI 182780 IM or placebo IM over 2 minutes on day 1. Patients undergo surgery between days 8 and 29.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 3,656 patients (1,828 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage I or II primary operable breast cancer

  * Surgery planned within next 1-4 weeks
* Hormone receptor status:

  * Estrogen receptor positive or unknown
  * No known estrogen receptor negative tumor
  * Unknown progesterone receptor status eligible

PATIENT CHARACTERISTICS:

Age:

* Any age

Sex:

* Female

Menopausal status:

* Premenopausal or postmenopausal

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* No bleeding diathesis not compatible with an IM depot injection

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception during and for 2-3 months after study
* No other prior or concurrent malignancy except adequately treated basal cell carcinoma of the skin or cancer of the uterine cervix
* No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 2 months since prior ICI 182780

Radiotherapy:

* No prior radiotherapy to primary tumor

Surgery:

* See Disease Characteristics

Other:

* No other concurrent preoperative therapy for breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-11; Primary Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J.H. van de Velde, MD, PhD, FRCS, FRCPS, Study Chair — Leiden University Medical Center; Anthony Howell, MD, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom